CLINICAL TRIAL: NCT06569485
Title: Phase 2 Study Evaluating Efficacy and Safety of Trilaciclib In Diffuse Large B-Cell Lymphoma Patients Receiving The Standard Chemotherapy R-CHOP.
Brief Title: A Study of Trilaciclib Combined With Chemotherapy in the Treatment of Diffuse Large B-Cell Lymphoma Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhiming, Chief Physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B2024-253-01
Record Dates: First submitted 2024-08-07; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: DLBCL

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention/Treatment (Experimental): Experimental: Trilaciclib+R-CHOP
  Patients with DLBCL were treated with Trilaciclib (240mg/m2, d1, within 4 hours before each chemotherapy) combined with Rituximab (375 mg/m2，d0), Cyclophosphamide (50 mg/m2，d1), Doxorubicin (50 mg/m2，d1) or Epirubicin（60 mg/m2，d1）, Vincristine (1.4 mg/m2), and Prednisone (100 mg，d1-5).
  A total of 6 cycles of treatment were performed every 21 days as a cycle.
  Interventions: Drug: Trilaciclib+R-CHOP

INTERVENTIONS:
Drug: Trilaciclib+R-CHOP — This is a prospective, single-arm, multi-center, phase II clinical study to evaluate the efficacy and safety of Trilaciclib in DLBCL patients treated with R-CHOP.
  Other Names: G1T28

SUMMARY:
This is a prospective, single-arm, multi-center, phase II clinical study to evaluate the efficacy and safety of Trilaciclib in DLBCL patients treated with R-CHOP.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center, phase II clinical study to investigate the myeloprotection efficacy, antitumor efficacy, and safety of Trilaciclib in DLBCL patients treated with R-CHOP (rituximab, cyclophosphamide, doxorubicin or Epirubicin, vincristine, and prednisone). 38 eligible subjects who met the inclusion criteria were screened and given a treatment regimen of Trilaciclib before chemotherapy R-CHOP, after signing informed consent. The incidence of Grade ≥ 3 neutropenia was used as the primary endpoint to observe whether Trilaciclib could reduce the occurrence or degree of chemotherapy-induced myelosuppression (CIM). Researchers will monitor potential adverse events (AEs) throughout the entire trial and grade the severity of adverse events according to the guidelines of the National Cancer Institute (NCI) Common Terminology for Adverse Events (CTCAE) 5.0.

ELIGIBILITY:
Inclusion Criteria:

1. Having sufficient understanding of this study and being willing to sign the informed consent form (ICF);
2. Age above 18 years old (including 18 years old)，regardless of gender;
3. Treatment-naive, histologically confirmed DLBCL, at least one tumor lesion that could be measured accurately at baseline according to RECIST1.1 criteria;
4. IPI score 0-2;
5. ECOG score of 0-2；
6. No prophylactic G-CSF, TPO, IL-11, ESA, iron within 1 week of screening hematology test, and no platelet transfusion or blood transfusion；
7. Estimated survival greater than 3 months；
8. Adequate organ function；
9. Being willing and able to comply with the visits, treatment plan, laboratory examinations and other study procedures scheduled in the study;
10. Women of childbearing potential must undergo a serum pregnancy test within 3 days prior to the first dose and the result must be negative. Female patients of childbearing potential and male subjects whose partners are women of childbearing potential must agree to use highly effective contraceptive methods during the study period and within 3 months after the last dose of study drug.

Exclusion Criteria:

1. The subject is participating in other interventional clinical studies;
2. The subject has previous or concurrent other malignancies;
3. Lymphoma bone marrow invasion;
4. The presence of symptomatic brain metastases requiring immediate radiotherapy or steroid therapy;
5. Known hypersensitivity to the applied drugs or any excipients；
6. Previous hematopoietic stem cell or bone marrow transplantation；
7. Active infection requiring systemic treatment;
8. Patients with uncontrolled cardiac clinical symptoms or diseases;
9. The subject has severe active infection or unexplained fever > 38.5 degrees during screening or before the first dose (the subject can be enrolled due to tumor fever as judged by the investigator);
10. Radiotherapy or radiotherapy at any site within 2 weeks before study medication;
11. Any investigational drug within 4 weeks before study medication;
12. Live attenuated vaccine within 4 weeks before study medication or possibly during the study period, influenza vaccine can be administered during the influenza season;
13. Pregnant or lactating women;
14. Any reasons that the investigator believes that it should be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Grade 3/4 neutropenia | Up to 6 months
  Proportion of subjects with at least one absolute neutrophil count (ANC) < 1.0 × 10^9/L enrolled and treated with at least one dose of trilaciclib

SECONDARY OUTCOMES:
ORR | Up to 6 months
  Objective Response Rate (ORR) is defined as the percentage of participants achieving complete response (CR) and partial response (PR) for tumor volume reduction and maintaining the minimum duration requirement based on RECIST v1.1
2y-PFS | Up to 2 years
  Progression-free survival (PFS per RECIST 1.1) is defined as the time until the first imaging disease progression or death (whichever occurs first)
2y-OS | Up to 2 years
  Overall survival (OS) is defined as the time until the subject's death due to any reason
Neutrophil-related myeloprotection efficacy | Up to 6 months
  Occurrence of febrile neutropenia adverse events(AEs)
Neutrophil-related myeloprotection efficacy | Up to 6 months
  Occurrence of Granulocyte colony-stimulating factor(G-CSF) administration
RBC related myeloprotection efficacy | Up to 6 months
  Occurrence of Grade 3/4 decrease of hemoglobin, occurrence and number of RBC transfusions on/after Week 5
RBC related myeloprotection efficacy | Up to 6 months
  Occurrence of erythropoiesis-stimulating agent(ESA) administration
Platelet related myeloprotection efficacy | Up to 6 months
  Occurrence of Grade 3/4 decrease of platelets
Platelet related myeloprotection efficacy | Up to 6 months
  Occurrence and number of platelet transfusions
Platelet related myeloprotection efficacy | Up to 6 months
  Occurrence of rhTPO/Recombinant human interleukin-11(rhIL-11) administration
Myeloprotection efficacy | Up to 6 months
  Hospitalization due to chemotherapy-induced myelosuppression
Chemotherapy dosing | Up to 6 months
  Chemotherapy dose reductions and delays due to chemotherapy-induced myelosuppression
Incidence of Treatment-Emergent Adverse Events | Up to 6 months
  To assess the effects of trilaciclib administered prior to chemotherapy on the occurrence and severity of adverse events by CTCAE 5.0, study treatment discontinuation due to adverse events, and trilaciclib adverse events of special interest.

OTHER OUTCOMES:
Exploratory analysis of potential biomarkers related with the outcome | Up to 6 months
  The change from baseline in immune cell levels in peripheral blood after treatment includes, but is not limited to:
  T cells (CD3, CD4, and CD8) B cells (CD19) Effector T cells (IFN-γ-producing CD4+ T cells, IL-2-producing CD4+ T cells, IL-17-producing CD4+ T cells, IFN-γ-producing CD8+ T cells, IL-2-producing CD8+ T cells) T cell activation markers (HLA-DR+ CD4+ T cells, HLA-DR+ CD8+ T cells) Regulatory T cells (Treg cells) (FoxP3, CD25, and CD127) Proportion of cells in the S phase
Exploratory analysis of potential biomarkers related with the outcome | Up to 6 months
  Tumor Biomarkers: Including but not limited to the relationship between the CDK4/6-Cyclin D-RB pathway and antitumor efficacy, the relationship between PD-L1, Ki67, and antitumor efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China